CLINICAL TRIAL: NCT05021328
Title: A Phase Ib Study on Toripalimab Combined With Anlotinib and SBRT for Patients With Untreated Brain Metastases of Driven Gene-negative Non-small Cell Lung Cancer
Brief Title: Toripalimab Combined With Anlotinib and SBRT in Patients With Untreated Brain Metastases of Driven Gene-negative NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Clinical Professor, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBCH-RT-2021-01
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: NSCLC
Keywords: Brain metastasis; Toripalimab; Anlotinib; SBRT; Drive gene negative
MeSH Terms: conditions — Brain Neoplasms | interventions — toripalimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib combined with SBRT (Experimental): Induction therapy (D1-D21): SBRT 7Gy✖️5 QD, D1-D5 + Anlotinib 12mg, QD, PO, D1-D14；
  Maintenance (D22~1year): Toripalimab 240mg iv drip D1 Q3W + Anlotinib 12mg, QD, PO, D1-D14, Q3W, until progression (up to approximately 1 year)
  Interventions: Drug: Anlotinib; Drug: SBRT 7Gy✖️5 QD
- Anlotinib combined with SBRT and Toripalimab (Experimental): Induction therapy (D1-D21): SBRT 7Gy✖️5 QD, D1-D5 + Toripalimab 240mg iv drip D1 + Anlotinib 12mg, QD, PO, D1-D14；
  Maintenance (D22~1year): Toripalimab 240mg iv drip D1 Q3W + Anlotinib 12mg, QD, PO, D1-D14, Q3W, until progression (up to approximately 1 year)
  Interventions: Drug: Toripalimab; Drug: Anlotinib; Drug: SBRT 7Gy✖️5 QD

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg, ivgtt, d1, q3w.
  Other Names: JS001; Toripalimab Injection; Teruipuli dankang Zhusheye; TuoYI
  Arms: Anlotinib combined with SBRT and Toripalimab
Drug: Anlotinib — Anlotinib 12 mg/d, d1-14, q3w.
  Other Names: AL3818; Anlotinib Hydrochloride Capsules; FuKeWei
Drug: SBRT 7Gy✖️5 QD — SBRT 7Gy✖️5 QD

SUMMARY:
The purpose of this study is to explore the efficacy and safety of toripalimab combined with anlotinib and SBRT for non-driver gene mutation untreated brain metastases non-small Cell Lung Cancer.

DETAILED DESCRIPTION:
Brain metastases (BM) develop in 22-54% of NSCLC patients during the disease course. NSCLC patients with BM with a median overall survival (OS) of 2-3 months when treated with systemic corticosteroid alone, and a median OS of 10-12 months when treated with brain radiation therapy. Recently, several studies have reported the benefits of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) for EGFR mutation NSCLC patients with BM. The median OS of EGFR mutation patients with BM significantly improved with TKIs treatment, which ranged from 11.8 to 18.8 months. However, for the EGFR wide-type NSCLC patients with BM, the prognosis remains poor.

JS-001 is the first monoclonal antibody (mAb) against programmed cell death protein-1 (PD-1) approved by the China Food and Drug Administration (CFDA) into the clinical trails.

Anlotinib hydrochloride is a multi-target receptor tyrosine kinase inhibitor that has significant inhibitory activity against angiogenesis related kinases such as VEGFR1/2/3, FGFR1/2/3, and other tumor related kinases such as PDGFR /, C-Kit, Ret, etc. (e.g., Met, FGFR1/2/3).

The previously study (2021 EMSO congress abstract) found that Apatinib, another kind of tyrosine kinase inhibitor that selectively inhibits the VEGFR-2, combined with brain radiation therapy could improve mOS time to 17 months in lung cancer patients with BMs.

Therefore, the investigators initiated this study to evaluate the efficacy and safety of toripalimab combined with anlotinib and SBRT for non-driver gene mutation untreated brain metastases non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender limit；
2. Pathologically or cytologically confirmed NSCLC, stage IV tumor with untreated BMs diagnosed by imaging 2 weeks before enrollment, 1~5 intracranial metastases (The primary tumor disease has not received systemic treatment, or brain metastasis occurs 6 months after the completion of postoperative adjuvant treatment or radical treatment);
3. Negative driver genes (EGFR, ALK, ROS1, etc.);
4. ECOG PS score: 0～1;
5. The expected survival time ≥ 3 months;
6. Intracranial metastases can be measured and evaluated by MRI;
7. Intracranial lesions are suitable for stereotactic radiotherapy based on the linear accelerator;
8. Able to independently complete neurocognitive tests;
9. Able to complete the QOL questionnaire independently;
10. Female subjects with fertility should undergo a urine or serum pregnancy test within 72 hours before receiving the first study drug administration, and prove to be negative, and are willing to use effectively during the test period to 3 months after the last administration Methods of contraception. For male subjects whose partners are women of childbearing age, effective methods of contraception should be used during the trial and within 3 months after the last administration;
11. The functions of important organs meet the following requirements (no blood components and cell growth factors are allowed to be used 2 weeks before the start of the research treatment): Absolute Neutrophil Count (ANC) ≥1.5×10 E+9/L, Hemoglobin (HB) ≥9g/dL, Platelets (PLT)≥90×10 E+9/L, Serum Albumin (ALB)≥2.8g/dL, Total Bilirubin (TBIL) ≤1.5 ULN, ALT、AST≤2.5 UILN(If abnormal liver function is caused by liver metastasis, ≤5 ULN), Serum creatinine sCr≤1.5 ULN, endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula) , Normal thyroid function;
12. The patients joined the study voluntarily and signed an informed consent form (ICF). They had good compliance and cooperated with follow-up.

Exclusion Criteria:

1. The lesion has received prior radiotherapy and is not suitable for SBRT;
2. Have leptomeningeal metastasis;
3. EGFR, ALK or ROS1 genomic tumour alterations;
4. Patients who cannot undergo MRI examination due to metal implants or claustrophobia;
5. Currently participating in interventional clinical research and treatment, or receiving other research drugs or treatment with research equipment within 4 weeks before the first administration;
6. Accept solid organ or blood system transplantation;
7. Past treatment history of CTLA-4, PD-1 or PD-L1 immune checkpoint inhibitors;
8. Has received VEGF pathway targeted therapy including anlotinib and bevacizumab.
9. Suffer from active autoimmune diseases that require hormone or immunomodulatory treatment, such as rheumatoid arthritis, ankylosing spondylitis, type I diabetes, psoriasis, vitiligo, immune-related thyroid dysfunction, etc. (hormone replacement Can be included after treatment is normal);
10. Suffer from acute or chronic infectious diseases, such as hepatitis B, hepatitis C, tuberculosis, and HIV;
11. Allergic to research drug ingredients
12. Active infection or fever of unknown cause occurred during the screening period and before the first administration> 38.5℃ (according to the judgment of the investigator, the subject can be included in the group due to fever caused by the tumor);
13. Suffer from uncontrolled clinical symptoms or diseases of the heart, such as:(1) Heart failure above NYHA II; (2) Unstable angina pectoris; (3) Myocardial infarction occurred within 1 year; (4) Patients with clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
14. Suffer from high blood pressure and cannot be well controlled by antihypertensive medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
15. Abnormal blood coagulation function (INR>2.0, PT>16s), have a bleeding tendency or are receiving thrombolytic therapy, and allow preventive use of low-dose aspirin and low-molecular-weight heparin;
16. Obvious coughing up blood or hemoptysis of 10ml or more per day in the 2 months before enrollment;
17. Have significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before enrollment;
18. Have received anti-tumor monoclonal antibodies (mAb) within 4 weeks before using the study drug for the first time, or the adverse events caused by the previously received drug have not recovered (ie ≤ grade 1 or reached the baseline level). Note: Except for subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 hair loss, if the subject has undergone major surgery, the toxic reaction and/or complications caused by the surgical intervention must be fully recovered before starting treatment;
19. Live vaccines have been vaccinated within 4 weeks before the first use of the study drug. Inactivated virus vaccines for seasonal influenza and injections are allowed, but live attenuated influenza vaccines for nasal use are not allowed;
20. The investigator judged other situations not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events | up to 24 month
  AEs per Common Terminology Criteria for Adverse Events (CTCAE V5.0)
Intracranial response rate (iORR) | 4 weeks after Radiotherapy.
  Proportion of patients with a complete or partial response in intracranial metastases as measured using RECIST 1.1 criteria (modified for brain metastases - bm RECIST).

SECONDARY OUTCOMES:
Intracranial progression-free survival (iPFS) | Tumor assesment at 4 weeks and 12 weeks after radiotherapy, and then every 12 weeks, up to 24 months
  Defined as the time from randomisation to progression of intracranial disease or death from any cause.
Local Control Rate (LCR) | Tumor assesment at 4 weeks and 12 weeks after radiotherapy, and then every 12 weeks, up to 24 months
  Local recurrence is defined as the onset or progression of nodular contrast grafting within the resection cavity according to the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.
Overall survival (OS) | Tumor assesment at 4 weeks and 12 weeks after radiotherapy, and then every 12 weeks, up to 24 months
  Defined as the time from randomisation to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No